CLINICAL TRIAL: NCT05350670
Title: Effect of Perineal Massage Combined With Cold Compress in the Second Stage on the Delivery Outcome of Primipara
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2022-07-103
Record Dates: First submitted 2022-03-09; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Cold Compress
Keywords: the second labor; perineal laceration; perineal massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- perineal massage and cold compress group (Experimental)
  Interventions: Behavioral: Perineal massage and cold compress
- no intervention group (No Intervention)

INTERVENTIONS:
Behavioral: Perineal massage and cold compress — Using perineal massage and cold compress during the second stage of labor to observe the effect
  Arms: perineal massage and cold compress group

SUMMARY:
Objective: The aim of this study was to investigate the effect of perineal massage and cold compress in second stage on the delivery outcome of primipara.

Method: This interventional study included a total of 200 primipara hoping for natural birth. Patients were randomly divided into two groups, one group used routine labor, one group used cold compress and perineal massage. Record the time of second stage of labor, degree of perineal laceration, etc.

ELIGIBILITY:
Inclusion Criteria:

* want give birth naturally
* have well developed perineum

Exclusion Criteria:

* Abnormal fetal position and head basin
* Severe obstetric complications

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
the time of second stage of labor | until the end of the second stage of labor
  calculate the time taken for the second stage of labor
Degree of perineal laceration | about 30 minutes after the pregnant woman gives birth
  The degree of perineal laceration was judged according to the degree of perineal division table
Lateral perineal resection rate | until the end of the second stage of labor
  observe whether perineal lateral excision was performed during delivery
Hospitalization days | up to 2 weeks
  observe how long pregnant women stay in the hospital